CLINICAL TRIAL: NCT02588859
Title: A Non-Interventional, Multicentre, Prospective, Observational Study to Understand Usage and Effect of Saxagliptin as First Add-On After Metformin in Indian Type 2 Diabetes Patients. (ONTARGET-India)
Brief Title: Study to Understand Usage and Effect of Saxagliptin as First Add-On After Metformin in Indian Type 2 Diabetes Mellitus Patients
Acronym: ONTARGET-INDIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1680R00019
Record Dates: First submitted 2015-10-12; First posted 2015-10-28 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes
Keywords: T2DM, Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multicentre, non-interventional, prospective, observational study which would be conducted in India to understand the usage and effect of saxagliptin as first add-on therapy after metformin. The study will enroll Type 2 Diabetes Mellitus (T2DM) patients who were inadequately controlled with metformin alone and have been recently prescribed saxagliptin as an add-on to metformin.

DETAILED DESCRIPTION:
This is a multicentre, non-interventional, prospective, observational study which would be conducted in India to understand the usage and effect of saxagliptin as first add-on therapy after metformin. The study will enroll Type 2 Diabetes Mellitus (T2DM) patients who were inadequately controlled with metformin alone and have been recently (i.e. within past 15 days) prescribed saxagliptin as an add-on to metformin.

The Investigator/designee would get signed informed consent from potential subjects of the study. The patients who meet all inclusion and none of the exclusion criteria will be enrolled in the study. These patients will then be assigned a patient identification number for the study. The Investigator/designee will collect the information as per the study schedule. This will be considered as Visit 1 of the patients. The patients will be managed as per the routine clinical practice of the physician for their condition and this study will neither interfere/advise the Investigators/designee for any drug/medication to be prescribed to the patients nor prescribe any intervention to them.The enrolled patients would then be asked to visit their respective study sites after 3 months ( +7 days) for the Visit-2 of study.

Around 50 study centers throughout India will be selected with a goal of enrolling up to 1500 patients (approximately 30 subjects each per site). The study will be initiated after obtaining written approval of Independent/Institutional Ethics Committee and written Informed consent of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to provide informed consent.
2. Female or male patients aged 18 years or above.
3. Patients with known case of Type 2 diabetes mellitus.
4. Patients with inadequate glycaemic control taking metformin monotherapy (minimum dose of 500 mg OD) for at least 3 months.
5. Patients who have recently (last 15 days) been prescribed saxagliptin in addition to metformin.

Exclusion Criteria:

1. Patients with Type 1 diabetes mellitus.
2. Patients taking glucose lowering drugs apart from metformin or saxagliptin.
3. Any medical condition of the patient which in the opinion of Investigator would interfere with safe completion of the study.
4. Pregnant or lactating women.
5. Women of childbearing potential not ready to use an effective barrier contraceptive method during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes patients
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2016-12-26 (Actual)

PRIMARY OUTCOMES:
Medication usage in enrolled subjects | at 3 months
  By Frequency of subjects taking different doses of saxagliptin and metformin

SECONDARY OUTCOMES:
Reduction in HbA1C | baseline and at 3 months
  Compare the reduction in HbA1C levels from baseline to follow up visit with baseline HbA1C levels

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sanjay Kalra, MD, DM (Endocrinology), Study Chair — Bharti Research Institute of Diabetes & Endocrinology, Karnal; Dr Bhavesh P Kotak, FRCS, MS, D Orth, Study Director — AstraZeneca Pharma India Ltd
Locations (31):
- India (31):
  - Research Site, Nellure, Andhra Pradesh
  - Research Site, Visakhapatnam, Andhra Pradesh
  - Research Site, Guwahati, Assam
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Karnāl, Haryana
  - Research Site, Yamuna Nagar, Haryana
  - Research Site, Bangalore, Karnataka
  - Research Site, Trivandrum, Kerala
  - Research Site, Kochi, Kochi
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Amritsar, Punjab
  - Research Site, Chandigarh, Punjab
  - Research Site, Ludhiana, Punjab
  - Research Site, Jaipur, Rajasthan
  - Research Site, Udaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Madurai, Tamiladu
  - Research Site, Hyderabad, Telangana
  - Research Site, Hyderebad, Telangana
  - Research Site, Allahābād, Uttar Pradesh
  - Research Site, Kanpur, Uttar Pradesh
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Noida, Uttar Pradesh
  - Research Site, Kolkata, West Bengal
  - Research Site, New Delhi

REFERENCES:
- [Derived] Kalra S, Bajaj S, Unnikrishnan AG, Baruah MP, Sahay R, Hardik V, Kumar A. Therapeutic Experience of Saxagliptin as First Add-on after Metformin in Indian Type 2 Diabetes Patients: A Non-interventional, Prospective, Observational Study (ONTARGET-INDIA). Indian J Endocrinol Metab. 2019 May-Jun;23(3):312-317. doi: 10.4103/ijem.IJEM_56_19. PMID 31641633
- See also: D1680R00019_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4017&filename=D1680R00019_CSR_Synopsis.pdf